CLINICAL TRIAL: NCT01519999
Title: Colorectal Cancer Screening With Improved Shared Decision Making (CRCS-WISDM)
Brief Title: Colorectal Cancer Screening With Improved Shared Decision Making
Acronym: CRCS-WISDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Allina Health System (Other); Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HM14436; WISDM-106965 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2012-01-13; First posted 2012-01-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer Screening; Shared Decision Making
Keywords: Shared decision making; Ambulatory Care; Patient-Centered Care; Community-wide intervention; Intervention Study; Longitudinal Studies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shared Decision Making (Experimental)
  Interventions: Behavioral: Shared Decision Making for Colorectal Cancer Screening
- Comparison (control) (No Intervention)

INTERVENTIONS:
Behavioral: Shared Decision Making for Colorectal Cancer Screening — Age-eligible adults in the intervention communities will be exposed to the shared decision-making intervention when they are seen in the primary care clinics (N=all patients 50-75 years seen during the study period who are non-adherent to CRCS recommendation). Additionally, among patients with primary care visits scheduled one week or more before the visit, they will be randomized to receive either a mailed decision aid booklet or an informational flyer on shared decision making and CRCS prior to the visit. Patients with primary care visits scheduled less than one week prior to the visit will not be mailed materials in advance. The effect of the pre-visit materials on referral to SDM session and CRCS adherence between these groups will be compared. They will also be exposed to shared decision-making tools and resources available through the community-wide intervention activities.
  Other Names: CRCS-WISDM
  Arms: Shared Decision Making

SUMMARY:
The purpose of this study is to increase colorectal cancer screening by implementing a community-wide shared decision-making (SDM) intervention, which embeds shared decision making within clinical practice and also uses an extensive community engagement campaign. The investigators hypothesize that colorectal cancer screening adherence will be higher in the intervention group (participating communities) compared to the usual care control group (non-participating comparison communities).

DETAILED DESCRIPTION:
Clinical practice: All patients 50-75 years seen in the participating primary care clinics during the study period who are non-adherent to CRCS recommendation. This sample is anticipated to be N~50,000 patients.

Community engagement: Includes mailed questionnaires to age-eligible adults residing in intervention and comparison (control) communities (N=2150).

ELIGIBILITY:
Inclusion Criteria:

* 50 to 75 years of age
* Lives in or receives care in the selected intervention or comparison (control) communities
* Average-risk for colorectal cancer
* Non-adherent to CRCS recommendation
* English-speaking
* People who consent to participate

Exclusion Criteria:

* <50 years of age or >75 years of age
* Not living in or receiving care in the selected intervention or comparison communities
* High-risk for colorectal cancer
* Adherent to CRCS recommendation
* Non-English speaking
* People who do not consent to participate

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206721 (Actual)
Dates: Start 2012-05; Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Change in colorectal cancer screening adherence | Baseline up to 24 months post intervention initiation
  Colorectal cancer screening adherence will be defined as having screening according to the recommendations of the United States Preventive Services Task Force. Participants will be classified as screened per recommendations if they have had fecal occult blood testing in the last year, flexible sigmoidoscopy in the last five years, or colonoscopy in the last ten years. Participants will be classified as non-adherent if they have not had any of the modalities within the recommended timeframe.

SECONDARY OUTCOMES:
Decisional conflict | Baseline up to 24 months post intervention initiation
  A previously validated decisional conflict scale, will be used, which includes 16 items all measured on a 5-point Likert-type scale. (e.g. difficulty in decision making, certainty with a decision, demonstrated feeling of understanding about risks and benefits of a decision, and satisfaction with a decision). Responses will be coded so that higher responses represent greater decisional conflict.
Modality-specific colorectal cancer screening barriers | Baseline up to 24 months post intervention initiation
  A previously validated modality-specific colorectal cancer screening barrier instrument will be used. The FOBT-specific scale includes 19 questions relating to barriers for fecal occult blood test and the colonoscopy-specific scale includes 21 questions relating barriers to colonoscopy. All items are measured on a 5-point Likert-type scale, with 5 representing greater barrier endorsement.
Colorectal cancer screening-related confusion | Baseline up to 24 months post intervention initiation
  Colorectal cancer-related confusion will be measured using 9 items which will be coded on a scale from 1 to 5 where 5 represents greater confusion endorsement.
Patients' shared decision-making experience | Baseline up to 12 months post intervention initiation
  Patients will answer multiple questions relating to their experience with the implementation of shared decision-making and their interactions with clinical staff. Items will be measured on Likert-like scales and will be coded so that higher scale numbers reflect more endorsement of positive opinions and experiences.
Providers'/staff shared decision-making experience | Baseline up to 24 months post intervention initiation
  Providers and staff will answer multiple questions relating to their experience with the implementation of shared decision-making with their patients in clinical practice. Items will be measured on Likert-like scales and will be coded so that higher scale numbers reflect more endorsement of positive opinions and experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Resa M Jones, MPH, PhD, Principal Investigator — Virginia Commonwealth University and Temple University
Locations (1):
- Allina Health Systems - Commons, Minneapolis, Minnesota, United States